CLINICAL TRIAL: NCT03991507
Title: Prospective Cohort Study for PCOS Patients in Clinical Reproductive Medicine Management System/Electronic Medical Record Cohort Database (CCRM/EMRCD)
Brief Title: PCOS (Polycystic Ovarian Syndrome) Patients
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Yingpu Sun, Director of Reproductive Medical Center, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: RMCZZU-PCOS cohort study
Record Dates: First submitted 2019-06-13; First posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Health Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Prospective Cohort Study for PCOS Patients was set up to investigate the short- and long-term health consequences in Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, China.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) affects 8-13% of women. It is a multifaceted condition characterized by chronic anovulation and excess ovarian activity.

Since last decade, Clinical Reproductive Medicine Management System/Electronic Medical Record Cohort Database (CCRM/EMRCD) has been used in Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, and Henan Province Key Laboratory for Reproduction and Genetics. Information of patients (POI, PCOS, Endometriosis, azoospermia, ect) were recorded comprehensively. The current project plans to recruit PCOS participants in our center. Biological samples, questionnaires and short/long term health data will be collected. The study is aimed to provide evidence for PCOS prognosis.

ELIGIBILITY:
Inclusion Criteria:

* PCOS patients diagnosed with The Rotterdam diagnostic criteria.

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: PCOS patients diagnosed with The Rotterdam diagnostic criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2050-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Level of serum FSH (Follicle stimulating hormone) | From date of inclusion, assessed by each 12 month, up to 40 years
  mIU/mL
Level of serum LH (Luteinizing hormone) | From date of inclusion, assessed by each 12 month, up to 40 years
  mIU/mL
Level of T (Testosterone) | From date of inclusion, assessed by each 12 month, up to 40 years
  ng/ml

SECONDARY OUTCOMES:
Body Weight | From date of inclusion, assessed by each 12 month, up to 40 years
  Recorded in Kilograms
Height | From date of inclusion, assessed by each 12 month, up to 40 years
  Recorded in centimeters

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive Medical Center, First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China